CLINICAL TRIAL: NCT05576740
Title: Influence of Menstrual Cycle Stages on Physical Fitness in Female Athletes
Brief Title: Influence of Menstrual Cycle Stages on Female Athletes
Status: Completed | Type: Observational
Sponsor: Universitat Jaume I (Other)
Responsible Party: Principal Investigator, Paula Recacha Ponce, Investigador principal, Universitat Jaume I
Other Study IDs: CD/77/2020
Record Dates: First submitted 2022-10-06; First posted 2022-10-12 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Menstrual Cycle; Sports
Keywords: Menstrual cycle; Performance; Hormonal verification; Contraception
MeSH Terms: interventions — Restraint, Physical; Activities of Daily Living

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- natural cycle: In this group, women have a natural menstrual cycle, not intervened by exogenous hormones. The interventions performed in this group are the same as in the other groups.
  Interventions: Procedure: Determination of hormone level concentrations; Procedure: Jump height determination; Procedure: Grip strength determination; Procedure: Flexibility determination; Procedure: Indirect maximum oxygen consumption determination; Device: Sensory and pain threshold determination; Other: Physical and mental symptoms associated with the menstrual cycle; Device: Daily activity; Procedure: Biochemical parameters determination; Procedure: Blood count determination; Procedure: Body composition parameters determination; Procedure: Vital signs; Procedure: Urinary LH determination
- artificial cycle: In this group, women with an artificial menstrual cycle, i.e. women using hormonal contraception, oral or vaginal, are selected. The interventions carried out in this group are the same as in the other groups.
  Interventions: Procedure: Determination of hormone level concentrations; Procedure: Jump height determination; Procedure: Grip strength determination; Procedure: Flexibility determination; Procedure: Indirect maximum oxygen consumption determination; Device: Sensory and pain threshold determination; Other: Physical and mental symptoms associated with the menstrual cycle; Device: Daily activity; Procedure: Biochemical parameters determination; Procedure: Blood count determination; Procedure: Body composition parameters determination; Procedure: Vital signs; Other: Checking for correct use of contraceptive methods
- natural cycle with deficient luteal phase: In this group, women have a natural menstrual cycle, with a low progesterone level during the luteal phase, and are not intervened by exogenous hormones. The interventions performed in this group are the same as in the other groups.
  Interventions: Procedure: Determination of hormone level concentrations; Procedure: Jump height determination; Procedure: Grip strength determination; Procedure: Flexibility determination; Procedure: Indirect maximum oxygen consumption determination; Device: Sensory and pain threshold determination; Other: Physical and mental symptoms associated with the menstrual cycle; Device: Daily activity; Procedure: Biochemical parameters determination; Procedure: Blood count determination; Procedure: Body composition parameters determination; Procedure: Vital signs; Procedure: Urinary LH determination

INTERVENTIONS:
Procedure: Determination of hormone level concentrations — Determination of concentration of 17β-oestradiol (pg/mL), progesterone (ng/mL), LH (mUI/mL), FSH (mUI/mL), prolactin (ng/mL), total testosterone (ng/mL), free testosterone (pmol/L) sex hormone binding globulin (SHBG) (nmol/L), cortisol (μg/dL), T3 (ng/dL), T4 (mcg/dL), TSH (mcU/mL), basal insulin (mcUI/mL) during the early follicular phase, late follicular phase, and mid-luteal phase.
Procedure: Jump height determination — by Chronojump contact mat, determine five types of jump in centimeters: Squat jump without additional weight, Squat jump with 50% of body weight, Countermovement jump, Abalakov jump, and Drop jump, during the early follicular phase, late follicular phase, and mid-luteal phase.
Procedure: Grip strength determination — measuring of changes in muscle strength by handgrip dynamometer in the hand to be tested (handgrip test) during the early follicular phase, late follicular phase, and mid-luteal phase. Three attempts on each hand.
Procedure: Flexibility determination — measurement of changes in the range of motion of the hamstring musculature, by sit and reach test (cm), during the early follicular phase, late follicular phase, and mid-luteal phase. Three tries.
Procedure: Indirect maximum oxygen consumption determination — by the Course Navette test, the indirect oxygen consumption is calculated using the formula: VO2max = (6xFA) - 27,4 (FA = Speed of the last stage of the test completed. It takes place during the early follicular phase, late follicular phase, and mid-luteal phase.
Device: Sensory and pain threshold determination — by electrical muscle stimulator (Digitimer DS7A), during the early follicular phase, late follicular phase, and mid-luteal phase.
Other: Physical and mental symptoms associated with the menstrual cycle — By The Daily Record of Severity of Problems (DRSP) questionnaire, during a full menstrual cycle.
Device: Daily activity — by accelerometer (GENEActiv) during a full menstrual cylcle: Wrist-worn device measuring accelerations as a measure of daily activity, in cpm, counts per minute.
Procedure: Biochemical parameters determination — Determination of concentration of iron (μg/dL), ferritin (ng/mL), and transferrin (mg/dL), during the early follicular phase, late follicular phase, and mid-luteal phase.
Procedure: Blood count determination — Determination of concentration of hemoglobin (g/dL), red blood cells (10^6/μL), hematocrit (%), white blood cells (10^3/μl), platelets (10^3/μl), during the early follicular phase, late follicular phase, and mid-luteal phase.
Procedure: Body composition parameters determination — Determination of weight (kg), total body water (L), proteins (kg), minerals (kg), body fat mass (kg), body mass index (BMI) (kg/m2), basal metabolic rate (kcal) by Bioelectrical Impedance Analysis, during the early follicular phase, late follicular phase, and mid-luteal phase.
Procedure: Vital signs — Determination of blood pressure (mmHg) and heart rate (bpm) at baseline, one minute and three minutes after the Course Navette test
Other: Checking for correct use of contraceptive methods — Pre-test questions about possible forgetfulness or mishandling of the method
  Groups: artificial cycle
Procedure: Urinary LH determination — Urine LH test strips are performed from day 8 of the cycle until positive.
  Groups: natural cycle; natural cycle with deficient luteal phase

SUMMARY:
The influence of the menstrual cycle on women's sports performance is still uncertain. Research on this topic shows methodological biases. The aim of the study will be to determine whether the menstrual cycle affects women's physical fitness, measuring this in 3 differentiated stages of the cycle: the early follicular phase, late follicular phase, and luteal phase. For this purpose, a blood test will be carried out in each phase, with hormone determination (oestradiol and progesterone) and a haemogram to determine the existence of possible anemia. After the extraction and other complementary tests (measurement of vital signs, bioimpedance...) the woman will undergo 3 physical tests to compare the results in the 3 phases. A group of women taking hormonal contraception will also be included, performing the same interventions. To determine whether the woman is ovulating or not, urinary luteinizing hormone (LH) strips will be given to the women and they will have to take them from day 8 of the cycle. In addition, women will wear an accelerometer to monitor their daily activity and to be able to observe if there is an influence on this stage of the menstrual cycle.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria natural cycles group:

* Female sex
* Women between 18 and 40 years of age
* Women who are members of a federation and who compete in a sport doing at least 240 minutes of exercise per week.
* Women with regular menstrual cycles (between 23 and 38 days long).
* Women who have not taken hormonal contraceptives (HA) for 6 months or more.

Inclusion criteria artificial cycles group:

* Female sex
* Women between 18-40 years of age
* Women federated and competed in a sport doing at least 240 minutes of exercise per week.
* Long-term users of HA (minimum 6 months).

Exclusion Criteria:

Exclusion criteria group natural cycles:

* Refusal to participate in the study
* Sedentary women
* Women on HA currently or in the 6 months before the study
* Women with irregular menstrual cycles, less than 23 or more than 38 days in length
* Any existing metabolic disease or disorder
* Regular use of medications or dietary supplements that could affect the results
* Pregnancy or breastfeeding

Exclusion criteria artificial cycles group:

* Refusal to participate in the study
* Sedentary women
* Any existing metabolic disease or disorder
* Regular use of medications or dietary supplements that could affect the results
* Inability to manage contraception in a disciplined manner

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — In this case, the study is aimed at women as it investigates the influence of the menstrual cycle on sports performance.
Study Population: Women between 18 and 40 years old, with regular menstrual cycles, who practice sport regularly, proven by federation and competition in a sport, and confirming the completion of at least 240 minutes of physical activity per week. In the case of women with hormonal contraception, they must be with the established method (minimum 6 months with it).
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2022-03-16 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Change in 17β-oestradiol concentration (in pg/mL) | three times in a month
  concentration of 17β-oestradiol in pg/mL
Change in T4 concentration (in mcg/dL) | three times in a month
  concentration of T4 in mcg/dL
Change in T3 concentration (in ng/dL) | three times in a month
  concentration of T3 in ng/dL
Change in cortisol concentration (in μg/dL) | three times in a month
  concentration of cortisol in μg/dL
Change in TSH concentration (in mcUI/mL) | three times in a month
  concentration of thyroid-stimulating hormone (TSH) and basal insulin in mcUI/mL
Change in SHBG concentration (in nmol/L) | three times in a month
  concentration of sex hormone binding globulin (SHBG) in nmol/L
Change in free testosterone concentration (in pmol/L) | three times in a month
  Concentration of free testosterone in pmol/L
Change in progesterone concentration (in ng/mL) | three times in a month
  Concentration of progesterone, prolactin and total testosterone in ng/mL
Change in LH and FSH concentration (in mUI/mL) | three times in a month
  Concentration of luteinizing hormone (LH) and FSH (follicle stimulating hormone) in mUI/mL
Change from baseline jumping height | three times in a month
  Measuring of change in muscle power through Squat jump without additional weight, Squat jump with 50% of body weight, Countermovement jump, Abalakov jump, and Drop jump by Chronojump contact mat, in cm. Three tries on each jump.
Change from baseline grip strength | three times in a month
  measuring of changes in muscle strength by handgrip dynamometer in the hand to be tested (handgrip test). Three attempts on each hand.
Change from baseline flexibility | three times in a month
  measurement of changes in the range of motion of the hamstring musculature, by sit and reach test (cm). Three tries.
Change from baseline indirect maximum oxygen consumption | three times in a month
  by the Course Navette test
Change from baseline sensory and pain threshold | three times in a month
  by electrical muscle stimulator (Digitimer DS7A)
Change from baseline physical and mental symptoms associated with the menstrual cycle by The Daily Record of Severity of Problems questionnaire | Duration of a full menstrual cycle (approximately 28 days)
  By The Daily Record of Severity of Problems (DRSP) questionnaire. This scale measures symptoms subjectively from 1 to 6, where 1 corresponds to "not at all" and 6 corresponds to "extreme". The higher the score, the more severe the symptom is.
Change from baseline daily activity | Duration of a full menstrual cycle (approximately 28 days)
  by accelerometer (GENEActiv): Wrist-worn device measuring accelerations as a measure of daily activity, in cpm, counts per minute.

SECONDARY OUTCOMES:
Change in iron concentration (in μg/dL) | three times in a month
  concentration of iron in μg/dL
Change in transferrin concentration (in mg/dL) | three times in a month
  concentration of transferrin in mg/dL
Change in ferritin concentration (in ng/mL) | three times in a month
  concentration of ferritin in ng/mL
Change in hemoglobin concentration (in g/dL) | three times in a month
  concentration of hemoglobin in g/dL
Change in white blood cells and platelets concentration (in 10^3/μl) | three times in a month
  concentration of white blood cells and platelets in 10^3/μl
Change in hematocrit concentration (in %) | three times in a month
  concentration of hematocrit in %
Change in red blood cells concentration (in 10^6/μl) | three times in a month
  concentration of red blood cells in 10^6/μL
Change in weight, proteins, minerals and body fat mass in kg | three times in a month
  Weight, proteins, minerals and body fat mass in kg by Bioelectrical Impedance Analysis
Change in Body Mass Index (BMI) in kg/m2 | three times in a month
  Body Mass Index (BMI) in kg/m2 by Bioelectrical Impedance Analysis and measuring tape
Change in Basal metabolic rate in kcal | three times in a month
  Basal metabolic rate in kcal by Bioelectrical Impedance Analysis
Change in total body water in liters (L) | three times in a month
  total body water in liters (L) by Bioelectrical Impedance Analysis
Change in Blood pressure in mmHg | three times in a month
  Blood pressure (systolic and diastolic pressure) in mmHg at baseline, one minute and three minutes after the Course Navette test by blood pressure monitor
Change in heart rate in bpm | three times in a month
  Heart rate in bpm at baseline, one minute and three minutes after the Course Navette test by blood pressure monitor

CONTACTS AND LOCATIONS:
Overall Officials: Paula Recacha-Ponce, Midwife, Principal Investigator — Universitat Jaume I; Eladio Collado-Boira, Doctor, Study Director — Universitat Jaume I; Carlos Hernando-Domingo, Doctor, Study Director — Universitat Jaume I
Locations (1):
- Jaume I University, Castellon, Castellon, Spain

IPD SHARING:
Plan to Share IPD: Yes
The aim is to publish the results obtained in high impact journals.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: results are expected to be available from 2023 when the data will be analysed and the results published.The data will always be available for consultation.
Access Criteria: open acces